CLINICAL TRIAL: NCT05222425
Title: Treatment of Non-severe SARS-CoV-2 Outpatients With Herbal Compound Xagrotin, Phase 3
Brief Title: Treatment of Non-severe Covid-19 Outpatients With Xagrotin, Phase 3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biomad AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-022022-FA3XAG/NO
Record Dates: First submitted 2022-02-01; First posted 2022-02-03 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Sars-cov-2
Keywords: sars-cov-2
MeSH Terms: interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group (Experimental): Patients in the Treatment arm receive Xagrotin extract 2 grams three times a day in combination to the standard of care for sars-cov-2.
  Interventions: Drug: Xagrotin
- Control group (No Intervention): Patients in the Control arm received the standard of care for sars-cov-2.
- Placebo group (Placebo Comparator): Patients in the Treatment arm receive green tea 2 grams three times a day in combination to the standard of care for sars-cov-2.
  Interventions: Drug: Green tea

INTERVENTIONS:
Drug: Xagrotin — A herbal compound
  Arms: Treatment group
Drug: Green tea — Normal green tea
  Arms: Placebo group

SUMMARY:
This is an interventional, multi-center, randomized study. Adults with confirmed covid-19 disease not more than 10 days before enrollment date will be recruited (n=1000). Patients in same condition who get treated with standard of care will be randomly assigned to the control group (n=1000), and patients in same condition who get treated with standard of care will be randomly assigned to the placebo group (n=1000). The investigators analyze the effect of Xagrotin, and also investigate impact of different characteristics for instance gender, age, duration of disease, smoking habits and concomitant diseases on the outcome.

DETAILED DESCRIPTION:
An interventional, multi-center, randomized study that will performe in an outpatient setting (n=1000). Adults with confirmed covid-19 disease not more than 10 days before enrollment date will be recruited. Patients in same condition who had treated with standard of care will randomly assign to the control group (n=1000), and patients in same condition who get treated with standard of care will be randomly assigned to the placebo group (n=1000). The investigators analyze the effect of Xagrotin, and also investigate impact of different characteristics for instance gender, age, duration of disease, smoking habits and concomitant diseases on the outcome. Adverse events will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or higher
* Newly diagnosed (no longer than 10 days)
* PCR or clinically confirmed Covid-19

Exclusion Criteria:

* Coronavirus patients admitted to medical centers for hospitalization and receive medical treatment and necessary care in medical centers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-12-07 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  Number of Participants who die by day 30 after the enrollment

SECONDARY OUTCOMES:
Duration of Disease From Beginning of Treatment | 30 days
  Number of days the patient has experienced the symptoms
Hospitalization | 30 days
  Number of participants who have been hospitalized for Covid-19
Duration of Hospitalization When Occurred | 30 days
  Days the participants were hospitalized

CONTACTS AND LOCATIONS:
Locations (1):
- Directorate of health of Sulaimani, Iraq -KRG, Sulaymaniyah, Iraq

IPD SHARING:
Plan to Share IPD: No